CLINICAL TRIAL: NCT03085420
Title: Cardiac Arrhythmias and Dysfunction in the Pediatric Burn Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participating site withdrew prior to any enrollment and lead site with slow enrollment. Not expected to meet enrollment goals.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Ivan Wilmot, Principal Investigator, Shriners Hospitals for Children
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: CIN1604
Record Dates: First submitted 2017-01-19; First posted 2017-03-21 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Cardiac Dysfunction
Keywords: Burns; Pediatrics; Cardiac Arrhythmia
MeSH Terms: conditions — Burns; Arrhythmias, Cardiac | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ≥30% TBSA burn injury (Experimental): For patients in Group 1 with ≥30% TBSA, a baseline Echocardiogram (ECHO) will be obtained approximately one week from admission and monthly (+/- 1 week) or at an interval determined by cardiology during the acute inpatient stay. ECHO tests will be discontinued after 3 negative exams or when discontinued by cardiology, whichever comes first.
  Interventions: Diagnostic Test: Echocardiogram
- <30% TBSA burn injury (No Intervention): For patients in Group 2 with <30% TBSA and presence of a cardiac abnormality standard clinical care appropriate for the type of arrhythmia will be followed.

INTERVENTIONS:
Diagnostic Test: Echocardiogram — A baseline Echocardiogram test (ECHO) will be done one week from admission and monthly (+/- 1 week) or as ordered by a cardiologist.
  Other Names: ECHO
  Arms: ≥30% TBSA burn injury

SUMMARY:
The purpose of this study is to collect information about how often an abnormal heart beat happens in children who have been burned.

DETAILED DESCRIPTION:
The investigators hope to learn the following:

* If heart arrhythmias are more common in children with a large burn injury than in children with a small burn injury.
* The difference in development of a heart arrhythmia after a large burn injury by comparing information from children with large burns who do and do not develop a heart arrhythmia.
* A better understanding of the length of a hospital stay, the number of operations, and the number of care complications in patients with heart arrhythmias after a burn injury.

ELIGIBILITY:
Inclusion Criteria:

Pediatric burn patients from age 0 - 18 who have sustained a burn injury will be eligible for this study.

Group 1 will consist of patients with ≥30% TBSA burn injury. Group 2 will consist of patients with <30% TBSA burn injury who develop a cardiac abnormality.

Exclusion Criteria:

Patients with pre-existing cardiac disorder, desquamative skin disorders and electrical injury.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Frequency of cardiac dysfunction in pediatric burn patients | Through study completion up to 4 years after hospital discharge.
  Results of echocardiograms will be compared between patients with cardiac dysfunction versus those without cardiac dysfunction.

SECONDARY OUTCOMES:
Acute care hospital length of stay | Hospital admission to discharge (average of 1 day per %TBSA burn - example 30 days for a 30% TBSA burn injury).
  Hospital length of stay (admission date to discharge date) will be compared between participants with cardiac dysfunction versus participants without cardiac dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wilmot, MD, Principal Investigator — Shriners Hospitals for Children; Petra M Warner, MD, Study Director — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak GZ, Hardy AR, Meyer RA, Kagan RJ. Reversible cardiomyopathy after severe burn injury. J Burn Care Res. 2006 Jul-Aug;27(4):482-6. doi: 10.1097/01.BCR.0000226018.30433.ED. PMID 16819352
- [Background] Howard TS, Hermann DG, McQuitty AL, Woodson LC, Kramer GC, Herndon DN, Ford PM, Kinsky MP. Burn-induced cardiac dysfunction increases length of stay in pediatric burn patients. J Burn Care Res. 2013 Jul-Aug;34(4):413-9. doi: 10.1097/BCR.0b013e3182685e11. PMID 23237822
- [Background] Guillory AN, Clayton RP, Herndon DN, Finnerty CC. Cardiovascular Dysfunction Following Burn Injury: What We Have Learned from Rat and Mouse Models. Int J Mol Sci. 2016 Jan 2;17(1):53. doi: 10.3390/ijms17010053. PMID 26729111